CLINICAL TRIAL: NCT04423107
Title: Assessment of Postoperative Pain in Boys Undergoing Hypospadias Repair
Brief Title: Assessment of Postop Hypospadias Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypospadias Repair Project
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Hypospadias
Keywords: pediatric hypospadias repair
MeSH Terms: conditions — Hypospadias | interventions — Acetaminophen; Ibuprofen; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No opioid (Active Comparator): Acetaminophen every 6 hours and Ibuprofen every 6 hours
  Interventions: Drug: Acetaminophen, Ibuprofen
- Opioid (Active Comparator): Acetaminophen every 6 hours, Ibuprofen every 6 hours, and Oxycodone every 6 hours as needed for breakthrough pain for 10 doses.
  Interventions: Drug: Acetaminophen, Ibuprofen, Oxycodone

INTERVENTIONS:
Drug: Acetaminophen, Ibuprofen — Acetaminophen (Tylenol) 15 mg/kg q6h and Ibuprofen (10 mg/kg) q6h
  Other Names: Tylenol (Acetaminophen)
  Arms: No opioid
Drug: Acetaminophen, Ibuprofen, Oxycodone — Acetaminophen (Tylenol) 15 mg/kg q6h, Ibuprofen q6h, and Oxycodone 0.1 mg/kg q6h
  Other Names: Tylenol (Acetaminophen)
  Arms: Opioid

SUMMARY:
One of the most common pediatric urology procedures is hypospadias repair, a surgery to correct curvature of the penis and move the urethral meatus into the glans. A survey of pediatric urologists demonstrated that 72% of pediatric urologists prescribe opioid pain medication following the procedure. Using a validated questionnaire, the investigators aim to quantify how much opioid pain medication boys undergoing hypospadias repair require and if opioid pain medication can be eliminated from the routine postoperative medication regimen.

DETAILED DESCRIPTION:
Postoperative pain scores, as measured by the Parents' Postoperative Pain Measure scale, will not be statistically different in boys who receive opioid pain medication postoperatively compared to boys who do not.

The long-term objectives of this study are to understand if pre and postoperative counseling and education along with proper surgical technique will result in less opioid prescriptions following hypospadias repair.

Children with suspected hypospadias will be seen and examined in clinic and offered surgery if appropriate. If the families elect for surgery, this will be performed by one of the investigators between 6-12 months of age. The surgical technique may vary among the investigators. Patients with severe hypospadias may require multiple surgeries for correction.

On the day of surgery, patients will be randomized to receive one of two pain medication regimens:

1. Acetaminophen (15 mg/kg) q6h and Ibuprofen (10 mg/kg) q6h
2. Acetaminophen q6h, Ibuprofen q6h, and Oxycodone 0.1 mg/kg q6h prn breakthrough pain for 10 doses Home dosing regimens will be started six hours after the last hospital dose of each medication. The families will be instructed as to when they can give oral medications at home. Lastly, families of both children in both groups will be instructed to contact the clinic or urologist on call if their children are experiencing uncontrolled pain. This may necessitate evaluation in person or adjustment of the current pain regimen. Any deviation from to prescribed pain regimen will be recorded for the study.

Patients will be contacted by phone at 1, 3, and 5 days postoperatively and given a validated questionnaire, the Parents' Postoperative Pain Measure scale, to objectively quantify how much discomfort boys in both groups experienced.

ELIGIBILITY:
Inclusion Criteria:

All boys undergoing hypospadias repair at our institution between June 2020 and June 2021

Exclusion Criteria:

Boys who have a contraindication to caudal block or Acetaminophen, Ketorolac, Ibuprofen, or Oxycodone use. Boys over 2 years of age.

Ages: 6 Months to 23 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — All boys undergoing hypospadias repair at our institution
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of postop pain measured by Parents Postoperative Pain Measurement Scale | 1 year
  Assessment of postop pain as measured by Parents Postoperative Pain Measurement Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bhalaajee Meenakshi-Sundaram, MD, Principal Investigator — University of Oklahoma HSC, Dept. of Urology
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No